CLINICAL TRIAL: NCT02182063
Title: An Open Label Randomized Phase II Study of Oral Treatment With BIBF 1120 250 mg Twice Daily Versus 150 mg Twice Daily in Patients Suffering From Hormone Refractory Prostate Cancer After Progression With Docetaxel Based Regimen
Brief Title: A Study With BIBF 1120 in Patients With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.11
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — nintedanib

ARMS (2):
- BIBF 1120 low dose (Experimental)
  Interventions: Drug: BIBF 1120 low dose
- BIBF 1120 high dose (Experimental)
  Interventions: Drug: BIBF 1120 high dose

INTERVENTIONS:
Drug: BIBF 1120 low dose
  Arms: BIBF 1120 low dose
Drug: BIBF 1120 high dose
  Arms: BIBF 1120 high dose

SUMMARY:
The aim of this study was to evaluate the efficacy of two different doses of BIBF 1120 (250 mg twice daily versus 150 mg twice daily) in an exploratory manner. Safety, quality of life and pharmacokinetic parameters on a sub-sample of 20 patients were also analysed for the two different doses.

ELIGIBILITY:
Inclusion Criteria:

1. Patient written informed consent obtained prior to any study procedures and consistent with ICH-GCP (International Conference on Harmonization - Good Clinical Practice) guidelines and local law
2. Presence of histologically documented adenocarcinoma of the prostate
3. Presence of metastatic disease
4. Life expectancy of at least 3 months
5. Progression after orchidectomy or during LH-RH (Luteinising hormone - releasing hormone) analogs with castrate testosterone serum levels <30 ng/ml (chemical castration had to be continued) and absence of anti-androgen withdrawal syndrome
6. Minimum value of PSA = 20 ng/ml at screening
7. Stopping the previous treatment with docetaxel based regimen or/and with antiandrogen 4 weeks before the inclusion of the patient
8. ECOG performance status ≤ 2
9. Progression after only one previous chemotherapy with docetaxel based regimen:

   * Appearance of a new lesion or increase of an existing measurable / non measurable lesion
   * Increase of PSA ≥ 25% documented by two successive exams
   * Increase of pain if there is a correlation with a radiological progression or with a PSA increase as defined above
10. Adequate hepatic function: total bilirubin within normal limits, ALT (Alanine aminotransferase) and/or AST (aspartate aminotransferase) ≤ 1.5x upper limit of normal (ULN). Prothrombin time (PT) and partial thromboplastin time (PTT): maximum 50% deviation from normal limits
11. Adequate renal function: serum creatinine ≤ 2 x upper normal limit (UNL)
12. Absolute neutrophil count (ANC) ≥ 1500/mL, Platelets ≥ 100,000/mL, Hemoglobin ≥ 9.0 g/dL (hemoglobin may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors)

Exclusion Criteria:

1. Gastrointestinal disorders or abnormalities that would inhibit absorption of the study drug
2. Serious illness or concomitant non-oncological disease such as neurologic-, psychiatric-, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
3. Significant cardiovascular diseases (i.e. uncontrolled hypertension, instable angina, history of myocardial infarction or congestive heart failure >NYHA II (New York Heart Association) during the 6 previous months
4. Strontium or equivalent radioactive isotope during the 6 previous months
5. Concomitant second malignancy, with the exception of treated basal cell carcinoma of the skin or a recovered cancer at least since 5 years
6. Major injuries and surgeries within the past 4 weeks. Planned surgical procedures during the trial. Patients with incomplete wound healing
7. History of haemorrhagic or emerging thrombotic event. Known inherited predisposition to hemorrhage or thrombosis
8. Patients who require full-dose anticoagulation or heparinization or continuous treatment with acetylsalicyclic acid > 325 mg
9. Concomitant treatment with other experimental drugs or anti-cancer therapy including hormone therapy (except LH-RH agonists)
10. Biphosphonates during the study since four weeks prior to the inclusion of the patient
11. Known or suspected symptomatic brain metastases
12. Known or suspected symptomatic epiduritis
13. Treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy (visit 2) or concomitantly with this trial
14. Patients unable to comply with the protocol

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Decline of prostate specific antigen (PSA) of ≥20% | Up to week 25 after first drug administration

SECONDARY OUTCOMES:
Decline of prostate specific antigen (PSA) of ≥50% | Up to week 25 after first drug administration
Time to Tumour Progression (TTP) | Up to week 29
Incidence and intensity of Adverse Events | Up to week 34
Radiological response rate according RECIST (Response Evaluation Criteria in Solid Tumours) | Up to week 25 after first drug administration
Change in Eastern Cooperative Oncology Group (ECOG) performance status | Baseline, up to week 25
Duration of overall survival | Up to week 29 after first drug administration
Change in Prostate Specific Antigen Doubling Time (PSADT) | Baseline, up to week 25
Drug plasma concentration measurement | Up to week 23 after first drug administration
Change in Quality of Life (QoL) using the general questionnaire of the European Organization for Research and Treatment-Quality of Life Questionnaire (EORTC-QLQ-C30) | Baseline, up to week 25
Change in Pain Present Intensity (PPI) score | Baseline, up to week 25

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/24849708